CLINICAL TRIAL: NCT03040336
Title: Pilot Testing Prehabilitation Services Aimed at Improving Outcomes of Frail Veterans Following Major Abdominal Surgery
Brief Title: Piloting Prehabilitation Before Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PPO 16-335; HX-002345 (Other Grant/Funding Number: VA ORD HSR&D)
Record Dates: First submitted 2017-01-18; First posted 2017-02-02 (Estimated); Results first posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Frailty
Keywords: surgery; prehabilitation; exercise therapy; nutrition support
MeSH Terms: conditions — Frailty | interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prehabilitation (Experimental): Standard of care + Prehabilitation
  Interventions: Behavioral: Prehabilitation
- Standard of Care (No Intervention): Standard of Care

INTERVENTIONS:
Behavioral: Prehabilitation — The 6-week long prehabilitation intervention will include (1) strength and balance training; (2) inspiratory muscle training; and (3) nutritional coaching and supplementation.
  Arms: Prehabilitation

SUMMARY:
Frail Veterans are at increased risk for poor surgical outcomes, and as the Veteran population grows older and more frail, there is a critical need to identify effective strategies for reducing surgical risks for these patients. Prior research shows that inter-disciplinary rehabilitation strategies deployed after surgery enhance recovery and improve outcomes by building strength and improving nutrition. We believe that similar improvements may be obtained by using similar interventions before surgery to "prehabilitate" patients' capacity to tolerate the stress of surgery. The proposed research will examine the feasibility of a new, prehabilitation intervention aimed at improving postoperative surgical outcomes through preoperative exercise training and nutritional supplementation. Findings from the study will inform the design of a larger randomized controlled trial of the prehabilitation intervention. If proven effective, prehabilitation could benefit as many as 42,000 frail Veterans who are scheduled for major elective surgery each year.

DETAILED DESCRIPTION:
Background: Frail Veterans are at increased risk for poor surgical outcomes. Although surgeons operate safely on even the oldest old, if the elder is also frail, the stress of surgery can result in significant mortality, morbidity, and institutionalization. Frailty is a clinical syndrome marked by muscle atrophy, diminished strength, decreased physical activity, and exhaustion. It is independent of any specific disease, but it increases with age, and is a more powerful predictor of increased perioperative mortality, morbidity, length of stay, and cost than predictions based on age or comorbidity alone. As the Veteran and US populations grow older and more frail, it is critically important to identify effective strategies for improving the surgical outcomes of these patients.

"Prehabilitation" has the potential to improve surgical outcomes among the frail. Prior research demonstrates that inter-disciplinary rehabilitation strategies deployed after surgery enhance recovery and improve outcomes by building strength, improving nutrition, and optimizing home supports. Based on this success, there is growing interest in deploying similar interventions before surgery in what some call "prehabilitation." By modifying physiological and environmental risks, prehabilitation aims to augment patients' capacity to compensate for the stress of both surgery and recovery. Frail patients will likely benefit disproportionately from prehabilitation because they have the most diminished capacity to adapt to the stress of surgery. However, prehabilitation has not yet been studied in either Veteran or specifically frail populations.

Objectives: We will examine the feasibility of a novel, multifaceted pre-habilitation intervention aimed at improving postoperative outcomes for frail Veterans undergoing major abdominal surgery. Specific aims are to:

1. Estimate rates of recruitment, randomization, retention, and compliance with the prehabilitation intervention;
2. Measure (a) physical performance, (b) pulmonary function, and (c) nutrition at baseline and 2-week intervals to estimate changes over time and explore the optimal duration of prehabilitation (2 vs. 4 vs. 6 weeks); and
3. Estimate overall and treatment-specific summary statistics for postoperative outcomes in terms of 30- and 90-day (a) mortality, (b) major complications, (c) length of hospital stay, (d) health-related quality of life, (e) quality of surgical care, and (f) change in level of independent living.

Methods: This randomized pilot study will enroll a consecutive cohort of up to 50 Veterans identified as frail using a standardized frailty assessment and scheduled for major abdominal surgery on the general or urological surgery services at the VA Pittsburgh Healthcare System. We will randomize participants 1:1 to receive either: (1) standard preoperative optimization by the Interdisciplinary Medical Preoperative Assessment Consultation & Treatment Clinic (IMPACT), or (2) prehabilitation + standard IMPACT optimization. The 6-week long prehabilitation intervention will include (1) strength and balance training; (2) inspiratory muscle training; and (3) nutritional coaching and supplementation. Assessments will include standard postoperative outcomes as well as the Short Physical Performance Battery to measure physical performance, Maximal Inspiratory Pressure to measure pulmonary function, and both prealbumin and the 7-point Subjective Global Assessment to measure nutrition. Outcomes will be assessed 30 or 90 days after surgery. Compliance with the prehabilitation regimen will be assessed through patient logs and pedometers. Analyses will inform the development of a larger randomized controlled trial testing the prehabilitation intervention. Findings will be relevant for the as many as 42,000 frail Veterans scheduled for major elective surgery each year.

ELIGIBILITY:
Inclusion Criteria:

* Frail as defined by an Risk Analysis Index (RAI) score >=16
* Scheduled for Major Abdominal Surgery as defined by a procedure that plans to violate the peritoneum or retroperitoneum (excluding inguinal hernias)

Exclusion Criteria:

* Unable to participate in planned Prehabilitation regimen
* Surgery is cancelled by IMPACT clinic or surgeon due to unacceptable risk
* Left ventricular ejection fractions <35%
* Severe valvular heart disease
* Significant arrhythmia
* Cognitive impairments that necessitate surrogate informed consent for the planned surgery
* Unable to speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2018-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E. Hall, MD MDiv MHSc, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (1):
- VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: Patient received the standard hospital care
Period: Overall Study
Arm/Group | Prehabilitation | Standard of Care
Started | 10 | 7
Completed | 7 | 4
Not Completed | 3 | 3
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prehabilitation | Standard of Care | Total
Number analyzed (Participants) | 10 | 7 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 9 | 6 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.22 (7.48) | 71.71 (11.08) | 73.69 (7.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 7 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 7 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 8 | 5 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Rate
Description: Recruitment will be expressed as the percentage of eligible patients approached who agree to participate in this pilot study.
Time Frame: Baseline
Population: 54 is the number of patients approached. Only 17 were consented and overall analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Approached: Patients approached to participate.
Arm/Group | Approached
Number analyzed (Participants) | 54
Participants | 17

2. Primary Outcome: Randomization Rate
Description: Randomization rate will be expressed as the percentage of eligible patients who agreed to participate who then agreed to be randomized to control or intervention conditions
Time Frame: Baseline
Population: 17 participants were overall analyzed. 10 were randomized to prehab, 7 were randomized to standard of care.
Measure: Count of Participants; unit: Participants
Arm/Group | Prehabilitation | Standard of Care
Number analyzed (Participants) | 17 | 17
Participants | 10 | 7

3. Primary Outcome: Retention Rate
Description: Retention rate will be expressed as the percentage of enrolled patients who were retained in the study and completed study procedures. It will be calculated for incremental steps along the study timeline and at the completion of study procedures 90 days postoperatively.
Time Frame: Baseline to 90 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Prehabilitation | Standard of Care
Number analyzed (Participants) | 10 | 7
Participants | 7 | 4

4. Primary Outcome: Compliance Rate
Description: Compliance rates will be expressed as the percentage of total compliance with assigned pehab activities actually completed by patients as recorded in home exercise and nutrition logs and completion of on site exercise sessions.
Time Frame: Baseline to Day of Surgery
Population: The compliance rate is only calculated for the prehabilitation arm.
Measure: Mean (Standard Deviation); unit: percentage of completed activities
Arm/Group | Prehabilitation
Number analyzed (Participants) | 10
percentage of completed activities
  Home exercise log | 56 (42.74)
  Nutrition log | 10 (31.62)
  On site exercise sessions | 93.6 (7.60)

5. Secondary Outcome: Grip Strength
Description: Grip strength will be measured in kilograms of pressure using a Jamar grip dynamometer
Time Frame: Baseline, day of surgery, 90 days postoperatively
Population: All participants that completed the hand grip assessment were analyzed at each completed timepoint.
Measure: Mean (Standard Deviation); unit: kgf/cm2
Arm/Group | Prehabilitation | Standard of Care
Number analyzed (Participants) | 10 | 7
kgf/cm2
  Baseline: number analyzed (Participants) | 10 | 6
  Baseline | 26.38 (4.99) | 27.75 (11.19)
  Day of Surgery: number analyzed (Participants) | 9 | 3
  Day of Surgery | 29.00 (5.38) | 32.00 (13.88)
  90 days: number analyzed (Participants) | 6 | 4
  90 days | 23.75 (4.23) | 33.63 (11.28)

6. Secondary Outcome: Pulmonary Function
Description: Pulmonary function will be measured in terms of maximal inspiratory and expiratory pressures.
Time Frame: Baseline, day of surgery, 90 days postoperatively
Population: All participants that completed the pulmonary function assessments were analyzed at each completed timepoint.
Measure: Mean (Standard Deviation); unit: cm of water
Arm/Group | Prehabilitation | Standard of Care
Number analyzed (Participants) | 10 | 7
cm of water
  Baseline Max MIP: number analyzed (Participants) | 10 | 6
  Baseline Max MIP | 66.00 (27.20) | 79.33 (30.81)
  Day of Surgery Max MIP: number analyzed (Participants) | 9 | 3
  Day of Surgery Max MIP | 70.11 (29.75) | 90.00 (19.97)
  90 Day Max MIP: number analyzed (Participants) | 6 | 3
  90 Day Max MIP | 63.17 (32.00) | 100.00 (11.53)
  Baseline Max MEP: number analyzed (Participants) | 10 | 6
  Baseline Max MEP | 90.60 (34.97) | 114.67 (41.56)
  Day of Surgery Max MEP: number analyzed (Participants) | 9 | 3
  Day of Surgery Max MEP | 108.67 (35.22) | 112.33 (35.64)
  90 Day Max MEP: number analyzed (Participants) | 6 | 4
  90 Day Max MEP | 97.67 (30.50) | 102.75 (19.48)

7. Secondary Outcome: Serum Prealbumin
Description: Nutrition will be measured by serum prealbumin. Higher scores indicate greater levels of protein. Lower levels indicate the potential of inflammation.
Time Frame: Baseline, day of surgery, 90 days postoperatively
Population: All participants that completed the blood draw were analyzed at each completed timepoint. Additionally, there was an error in the lab when processing the blood samples, this caused many samples to be evaluated incorrectly. Only correctly analyzed labs were included in this analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Prehabilitation | Standard of Care
Number analyzed (Participants) | 9 | 4
mg/dL
  Baseline Prealbumin: number analyzed (Participants) | 6 | 2
  Baseline Prealbumin | 26.5 (4.93) | 29 (2.83)
  Day of Surgery Prealbumin: number analyzed (Participants) | 2 | 2
  Day of Surgery Prealbumin | 22.5 (6.36) | 25.5 (2.12)
  90 Day Prealbumin: number analyzed (Participants) | 5 | 1
  90 Day Prealbumin | 23.6 (8.44) | 22 (0)

8. Secondary Outcome: Gait Speed
Description: Gait speed will be measured by using a stopwatch to time how long the patient takes to walk 4 meters.
Time Frame: Baseline, day of surgery, 90 days postoperatively
Population: All participants that completed the gait speed assessment were analyzed at each completed timepoint.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Prehabilitation | Standard of Care
Number analyzed (Participants) | 10 | 7
m/s
  Baseline Gait Speed | 0.98 (0.30) | 1.54 (0.55)
  Day of Surgery Gait Speed: number analyzed (Participants) | 9 | 2
  Day of Surgery Gait Speed | 1.00 (0.17) | 1.07 (0.15)
  90 Day Gait Speed: number analyzed (Participants) | 7 | 3
  90 Day Gait Speed | 1.07 (0.40) | 1.21 (0.20)

9. Secondary Outcome: Short Physical Performance Battery (SPPB)
Description: This standardized outcome measure asks patients to complete several activities that are scored independently and then aggregated into an overall score ranging from 0-12. Higher scores indicate better physical performance.
Time Frame: Baseline, day of surgery, 90 days postoperatively
Population: All participants that completed the SPPB assessments were analyzed at each completed timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prehabilitation | Standard of Care
Number analyzed (Participants) | 10 | 7
score on a scale
  Baseline SPPB: number analyzed (Participants) | 9 | 5
  Baseline SPPB | 9.13 (2.30) | 10.6 (1.52)
  Day of Surgery SPPB: number analyzed (Participants) | 9 | 2
  Day of Surgery SPPB | 10.56 (0.88) | 11 (0)
  90 Day SPPB: number analyzed (Participants) | 5 | 4
  90 Day SPPB | 9.8 (1.79) | 10.75 (0.96)

10. Secondary Outcome: Risk Analysis Index of Frailty (RAI)_questionnaire
Description: This recently published frailty index is assessed by a clinician administered questionnaire. The score and reflects frailty-associated mortality risk ranging from 0-81. Higher scores indicate higher risk for post operative complications and other frailty-related outcomes.
Time Frame: Baseline, day of surgery, 90 days postoperatively
Population: All participants that completed the RAI assessment were analyzed at each completed timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prehabilitation | Standard of Care
Number analyzed (Participants) | 10 | 7
score on a scale
  Baseline RAI: number analyzed (Participants) | 7 | 7
  Baseline RAI | 31.57 (11.86) | 24.75 (0.50)
  Day of Surgery RAI: number analyzed (Participants) | 7 | 2
  Day of Surgery RAI | 27.86 (12.79) | 29.00 (5.66)
  90 Day RAI: number analyzed (Participants) | 7 | 3
  90 Day RAI | 29.00 (10.39) | 26.67 (2.89)

11. Secondary Outcome: 7-point Subjective Global Assessment of Nutrition_questionnaire
Description: This standardized survey instrument is completed by a trained clinician after assessing a nutrition-specific patient history. The minimum score is 1 and the maximum score is 7. High scores indicate better nourishment.
Time Frame: Baseline, day of surgery, 90 days postoperatively
Population: All participants that completed the Subjective Global Assessment were analyzed at each completed timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prehabilitation | Standard of Care
Number analyzed (Participants) | 10 | 7
score on a scale
  Baseline Subjective Global Assessment: number analyzed (Participants) | 7 | 5
  Baseline Subjective Global Assessment | 5.43 (0.79) | 6.4 (0.55)
  Day of Surgery Subjective Global Assessment: number analyzed (Participants) | 7 | 4
  Day of Surgery Subjective Global Assessment | 5.14 (1.07) | 6.00 (0)
  90 Day Subjective Global Assessment: number analyzed (Participants) | 7 | 3
  90 Day Subjective Global Assessment | 5.14 (1.07) | 6.33 (0.58)

12. Other Pre Specified Outcome: Postoperative Mortality
Description: Postoperative mortality
Time Frame: 30 and 90 days postoperatively
Population: The mortality questionnaire was completed for all participants still enrolled in the study at the indicated time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Prehabilitation | Standard of Care
Number analyzed (Participants) | 9 | 4
Participants
  30-days mortality | 0 | 0
  90-days mortality: number analyzed (Participants) | 8 | 4
  90-days mortality | 1 | 0

13. Other Pre Specified Outcome: Health Related Quality of Life
Description: Assessment of Quality of Life (AQoL-6D). Utility score ranges from 0 to 1. Higher scores indicate better quality of life.
Time Frame: Baseline, day of surgery, 90-days postoperatively
Population: Not all participants were analyzed, because this measure requires participants to complete the questionnaire and not all participants did.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prehabilitation | Standard of Care
Number analyzed (Participants) | 7 | 3
score on a scale
  Baseline: number analyzed (Participants) | 7 | 2
  Baseline | 0.72 (0.09) | 0.67 (0.05)
  Day of Surgery: number analyzed (Participants) | 6 | 2
  Day of Surgery | 0.68 (0.08) | 0.77 (0.01)
  90-days postoperative: number analyzed (Participants) | 6 | 3
  90-days postoperative | 0.75 (0.09) | 0.80 (0.07)

14. Other Pre Specified Outcome: Quality of Surgical Care
Description: AHRQ Surgical Care Survey (SCS). Scores on this scale range from 1 to 3. Lower scores indicate better communication.
Time Frame: Day of Surgery and 30-days postoperatively
Population: All participants that completed the assessment were analyzed at each completed timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prehabilitation | Standard of Care
Number analyzed (Participants) | 9 | 5
score on a scale
  Day of Surgery Total Communication | 1.33 (0.37) | 1.13 (0.18)
  30-days Total Communication: number analyzed (Participants) | 7 | 4
  30-days Total Communication | 1.25 (0.29) | 1.19 (0.24)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each participant, from the time of enrollment, usually 3-6 weeks prior to surgery, to first final follow up, 90 days after surgery. Adverse events were collected over a time period of approximately four months.
Arm/Group | Prehabilitation | Standard of Care
All-Cause Mortality (participants affected / at risk) | 1/10 | 0/7
Serious Adverse Events (participants affected / at risk) | 3/10 | 2/7
Other Adverse Events (participants affected / at risk) | 0/10 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prehabilitation (N=10) | Standard of Care (N=7)
Unexpected and unrelated hospitalization (Injury, poisoning and procedural complications) | 3 (6) | 2 (2)
Unexpected and unrelated death (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Death due to prior diagnosis of lung cancer.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/36/NCT03040336/Prot_SAP_000.pdf